CLINICAL TRIAL: NCT02991937
Title: Comparison of Medical and Surgical Treatment of Uncomplicated Acute Appendicitis in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-00655
Record Dates: First submitted 2016-12-05; First posted 2016-12-14 (Estimated); Results first posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Piperacillin, Tazobactam Drug Combination; Surgical Procedures, Operative; Appendectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical Therapy (Active Comparator): Subjects in the medical therapy arm will be treated with piperacillin/tazobactam for at least 24 hours. Ciprofloxacin/metronidazole will be used in penicillin-allergic patients. Subjects will be maintained on nothing by mouth with intravenous fluids for at least 12 hours. Subjects will be transitioned to oral antibiotics when their WBC is normal, they have a decrease in CRP by ≥ 15%, and they have been afebrile for 24 hours on IV antibiotics.
  Interventions: Drug: Piperacillin/Tazobactam
- Surgical Intervention (Active Comparator): Subjects in the surgical treatment arm will receive intravenous antibiotics until the time of operation, and will be maintained on intravenous fluids and no oral intake until they undergo appendectomy as per standard of care. Appendectomy will occur within 24 hours of enrollment. Subjects in the surgical treatment arm will receive post-operative antibiotics as per standard of care.
  Interventions: Drug: Piperacillin/Tazobactam; Procedure: Surgical Treatment

INTERVENTIONS:
Drug: Piperacillin/Tazobactam — 24 hours of IV antibiotic administration
Procedure: Surgical Treatment — Appendectomy
  Other Names: Appendectomy
  Arms: Surgical Intervention

SUMMARY:
Several prior studies have demonstrated that medical management of acute appendicitis in adults is a safe first-line therapy option. This study aims to determine whether non-operative management of uncomplicated acute appendicitis with antibiotics is non-inferior to operative management in a pediatric population. This study will be a randomized controlled trial comparing non-operative management with antibiotics to surgical management of uncomplicated acute appendicitis. The hypothesis is that antibiotics are not worse than surgery for the treatment of uncomplicated appendicitis in children.

ELIGIBILITY:
Inclusion Criteria:

* first episode of appendicitis
* Pain < 48 hours
* White blood cell count < 18,000
* temperature < 103º F
* radiographic evidence of acute appendicitis on ultrasound or CT without evidence of perforation
* appendiceal diameter < 11 mm
* ability to take oral antibiotics

Exclusion Criteria:

* Prior antibiotic treatment for appendicitis
* presence of medical condition prohibiting surgical therapy
* radiographic or clinical evidence of abscess or perforation
* appendiceal mass, positive pregnancy test
* other diagnosis equally as likely as appendicitis
* pain for ≥ 48 hours, white blood cell count ≥ 18,000, temperature ≥ 103º F, or appendiceal diameter ≥ 11 mm
* inability to take oral antibiotics.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Fisher, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medical Therapy | Surgical Intervention
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medical Therapy | Surgical Intervention | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10.2 [8.5 to 11] | 9.7 [7.3 to 14.4] | 10 [8.4 to 11.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 14 | 13 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 9 | 20
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale - Parent
Description: Brief, standardized, generic assessment instrument that systematically assesses patients' and parents' perceptions of health-related quality of life (HRQOL) in pediatric patients with chronic health conditions using pediatric cancer as an exemplary model. PedsQL consists of 23 items scored on a 5-point Likert scale (0=never to 4=almost always). Items are reversed scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, and 4=0). The total score range is 0-100; the higher the score, the better the HRQOL.
Time Frame: 1 Year
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Medical Therapy | Surgical Intervention
Number analyzed (Participants) | 20 | 16
score on a scale | 91.3 [82.6 to 98.9] | 90.2 [70.1 to 97.0]

2. Secondary Outcome: Readmission Rates
Description: Percentage of patients readmitted to the hospital after discharge.
Time Frame: 1 Year
Measure: Number; unit: percentage of participants
Arm/Group | Medical Therapy | Surgical Intervention
Number analyzed (Participants) | 20 | 19
percentage of participants | 25 | 0

3. Secondary Outcome: Incidence of Long-term Complications in Medical Therapy Group
Description: Incidence of long-term complications will be reported as number of cases where appendicitis reoccurred resulting in appendectomies in participants of the medical therapy arm. This data will be obtained from medical record review.
Time Frame: 1 Year
Measure: Number; unit: Number of cases in 20 participants
Arm/Group | Medical Therapy
Number analyzed (Participants) | 20
Number of cases in 20 participants | 30

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Medical Therapy | Surgical Intervention
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 8/20 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medical Therapy (N=20) | Surgical Intervention (N=19)
Failure of Medical Therapy Requiring Surgery (Surgical and medical procedures) | 6 | 0
Readmission (Gastrointestinal disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT02991937/Prot_SAP_000.pdf